CLINICAL TRIAL: NCT05827081
Title: A Phase IIIb Study to Characterize the Efficacy and Safety of Adjuvant Ribociclib Plus Endocrine Therapy in a Close-to-clinical Practice Patient Population With HR+ HER2- Early Breast Cancer (Adjuvant WIDER)
Brief Title: Phase IIIb Study of Ribociclib + ET in Early Breast Cancer
Acronym: Adjuvant WIDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011O12001; 2022-503001-38-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Early Breast Cancer
Keywords: Hormone receptor positive (HR+); Human epidermal growth factor receptor-2 negative (HER2-); Early breast cancer (EBC); premenopausal; postmenopausal; male breast cancer; ribociclib; LEE011; Endocrine therapy (ET)
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — ribociclib; Letrozole; Goserelin; Leuprolide; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ribociclib + endocrine therapy (Experimental): Participants will receive ribociclib 400 mg orally once daily on days 1 to 21 of a 28-day cycle, in combination with daily endocrine therapy (ET) for 36 months (approximately 39 cycles). ET consists of:
  * For postmenopausal women: letrozole 2.5 mg orally once daily continuously, anastrozole 1 mg orally once daily continuously, or exemestane 25 mg once daily continuously.
  * For pre/perimenopausal women, and men: letrozole 2.5 mg orally once daily continuously, anastrozole 1 mg orally once daily continuously, or exemestane 25 mg once daily continuously, combined with goserelin subcutaneously (at 3.6 mg once every 4 weeks if the one-month depot formulation is used or at 10.8 mg once every 3 months if the three-month depot formulation is used) or leuprolide subcutaneously (at 3.75 mg once every 4 weeks if the one-month depot formulation is used or at 11.25 mg once every 3 months if the three-month depot formulation is used)
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Ansastrozole; Drug: Goserelin; Drug: Leuprolide; Drug: Exemestane

INTERVENTIONS:
Drug: Ribociclib — Ribociclib 400 mg orally once daily on days 1-21 of a 28 day cycle followed by 7 days rest
  Other Names: LEE011
Drug: Letrozole — Letrozole 2.5 mg orally once daily continuously
Drug: Ansastrozole — Anastrozole 1 mg orally once daily continuously.
Drug: Goserelin — Goserelin administered subcutaneously at 3.6 mg once every 4 weeks if the one-month depot formulation is used or at 10.8 mg once every 3 months if the three-month depot formulation is used
Drug: Leuprolide — Leuprolide administered subcutaneously at 3.75 mg once every 4 weeks if the one-month depot formulation is used or at 11.25 mg once every 3 months if the three-month depot formulation is used
Drug: Exemestane — Exemestane 25 mg once daily continuously

SUMMARY:
The purpose of this open-label, multicenter, phase IIIb, single-arm study is to characterize the efficacy and safety of the combination of ribociclib and standard adjuvant endocrine therapy (ET) on invasive breast cancer-free survival (iBCFS), in a close to clinical practice patient population with HR-positive (HR+), HER2-negative (HER2-), Anatomic Stage Group III, IIB, and a subset of Stage IIA Early Breast Cancer (EBC).

DETAILED DESCRIPTION:
The study consists of Screening, Treatment, and Follow-up periods.

* Treatment Period: all participants who complete screening will receive ribociclib 400 mg orally once daily on days 1 to 21 of a 28-day cycle, in combination with daily ET for 36 months (approximately 39 cycles) from the date of first dose. The Treatment Period starts when the patient receives their first dose of ribociclib and ends at the time of the 30-day Safety Follow-up. All treated participants should have a Safety Follow-up call conducted 30 days after the last dose of study treatment.
* Follow-up period: participants will be followed from 30 days after study treatment (i.e., ribociclib) completion/discontinuation (i.e. 30-day Safety Follow-up) until death, withdrawal of consent, lost to follow-up, or until 48 months after the last participant has received their first dose of study treatment (i.e. End of Study [EOS]), whichever occurs first.

ELIGIBILITY:
Key Inclusion criteria:

* Participant is an adult, male or female ≥ 18 years of age at the time of informed consent form signature (IC).
* Participant has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer (BC) based on the most recently analyzed tissue sample tested by a local laboratory prior to enrollment.
* Participant has HER2- BC defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing based on the most recently analyzed tissue sample.
* Participants may have already received any standard neoadjuvant and/or adjuvant ET, including tamoxifen or toremifene at the time of informed consent signature, but enrollment should occur within 36 months of prior ET start date and participants should have at least 3 years remaining of endocrine adjuvant therapy.
* For participants with prior ET treatment > 12 months, restaging is highly recommended (unless contradictory to local regulations) to rule out disease recurrence prior to enrollment.
* The number of participants with prior ET between 12 and 36 months will be capped at 30%. The cap will not apply to Black or African American participants.
* Participant has no contraindication to receive adjuvant ET in the study.
* Participant after surgical resection where tumor was removed completely, with the final surgical specimen microscopic margins free from tumor, and belongs to one of the following categories:

  * Anatomic Stage Group III, or
  * Anatomic Stage Group IIB, or
  * A subset of Anatomic Stage Group IIA.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Participant has adequate bone marrow and organ function.
* ECG values assessed by KardiaMobile-6L device, or standard 12-lead ECG per local investigator where KardiaMobile-6L cannot be used, as:

  * QTcF interval at Screening < 450 msec (QT interval using Fridericia's correction).
  * Mean resting heart rate 50-99 beats per minute (determined from the ECG).

Key Exclusion criteria:

* Participant with distant metastases of BC beyond regional lymph nodes (Stage IV according to AJCC 8th edition) and/or evidence of recurrence after curative surgery.
* Participant is concurrently using other antineoplastic therapy with the exception of adjuvant ET.
* Participant has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate participant participation in the clinical study or compromise compliance with the protocol, or limit life expectancy to ≤5 years.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial.
* Women of child-bearing potential (CBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 21 days after stopping the treatment.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2029-09-07 (Estimated); Study Completion 2030-09-20 (Estimated)

PRIMARY OUTCOMES:
Invasive Breast Cancer Free Survival (iBCFS) rate at 3 years | At 3 years
  iBCFS is defined as the time from the date of first dose to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), or contralateral invasive BC. iBCFS will be assessed using STEEP criteria version 2.0 (Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials), as assessed by Investigator.
  The iBCFS rate at 3 years will be assessed.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) using CTCAE v4.03 | Up to approximately 6 years
  To evaluate Safety of ribociclib + ET
Invasive Disease-Free Survival (iDFS) | Up to approximately 6 years
  iDFS is defined as the time from the date of first dose of study treatment to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), contralateral invasive BC, or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin). iDFS will be assessed using STEEP 2.0 as assessed by the investigator.
Distant Disease-Free Survival (DDFS) | Up to approximately 6 years
  Distant Disease-Free Survival (DDFS) is defined as the time from the date of first dose of study treatment to the date of the first event of recurrence at a distant site, death (any cause), or second primary non-breast invasive cancer (excluding in situ/non-invasive cancers and basal and squamous cell carcinomas of the skin).
  DDFS will be assessed using STEEP 2.0 as assessed by the investigator.
Distant Relapse-Free Survival (DRFS) | Up to approximately 6 years
  Distant Relapse Free Survival (DRFS) is defined as the time from the date of first dose of study treatment to the date of the first event of recurrence at a distant site or death (any cause). DRFS will be assessed using STEEP 2.0 as assessed by the investigator.
Recurrence-Free Interval (RFI) | Up to approximately 6 years
  RFI is defined as the time from date of first dose to date of first event of invasive recurrence in the ipsilateral breast or locoregionally, at a distant site, or death from breast cancer. RFI will be assessed using STEEP 2.0 as per investigator assessment.
Relative dose intensity (RDI) of ribociclib | Up to 3 years
  RDI is defined as the ratio of the dose intensity delivered to the planned dose intensity.
Overall Survival (OS) | Up to approximately 6 years
  OS is defined as time from the start of study treatment to date of death due to any cause.
Time To Discontinuation (TTD) of ribociclib | Up to 3 years
  TTD is defined as the time from starting ribociclib to the time to treatment discontinuation due to any cause.
Changes from baseline in Functional Assessment of Cancer Therapy - Breast (FACT-B) score | Up to approximately 6 years
  The FACT-B is a questionnaire that consists of 37 items with items from FACT-General (FACT-G) questionnaire (27 items) and from the Breast Cancer Subscale (BCS, 10 items). FACT-B consists of five subscales that address different aspects of the participant's quality of life: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and BCS.
Changes from baseline in Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) score | Up to approximately 6 years
  The FACT-ES is a questionnaire that consists of 19 items which assesses endocrine complaints and adverse events.
Changes from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score | Up to approximately 6 years
  The FACIT-F is a 13-item questionnaire designed to assess self-reported fatigue and its impact on daily activities and functions.
Changes from baseline in European Quality of Life-5 Dimensions (EQ-5D-5L) score | Up to approximately 6 years
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D-5L health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Changes from baseline in Work Productivity and Activity Impairment Questionnaire (WPAI-GH) score | Up to approximately 6 years
  WPAI-GH measures the impact of health problems on the participant's productivity, in paid or unpaid activities, in the last 7 days. It is 6-item scale measuring absenteeism, presenteeism, and impairments in unpaid activity.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (168):
- United States (58):
  - Central Alabama Research, Birmingham, Alabama
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Western Reg MC-COH Phoenix, Goodyear, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - Onco Inst of Hope and Innovation, Cerritos, California
  - City of Hope National Medical, Duarte, California
  - Providence Medical Foundation, Fullerton, California
  - Palo Alto Medical Foundation, Mountain View, California
  - UC Irvine Medical Center, Orange, California
  - Sutter Inst Medical Research, Sacramento, California
  - School Of Medicine, Sacramento, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Health, Fort Lauderdale, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Summit Cancer Care PC, Savannah, Georgia
  - Affiliated Oncologists IL, Chicago, Illinois
  - Hope And Healing Care, Hinsdale, Illinois
  - Midwestern Reg MC COH Chicago, Zion, Illinois
  - Investigative Clinical R of Indiana, Indianapolis, Indiana
  - University of Iowa Health Care, Waukee, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Minnesota Oncology Hematology P A, Minneapolis, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - HCA Midwest Division, Kansas City, Missouri
  - WA Uni School Of Med, St Louis, Missouri
  - Intermountain Healthcare, Billings, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Summit Health, Florham Park, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Presbyterian Medical Group, Albuquerque, New Mexico
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Clinical Research Alliance, Lake Success, New York
  - Mount Sinai School of Medicine, New York, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Oncology Associates of Oregon PC, Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Oregon Oncology Specialists Salem, Salem, Oregon
  - Consultants In Med Onco And Hema, Drexel Hill, Pennsylvania
  - Univ of Pittsburg Med Ctr Pinnacle, Harrisburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - El Paso Texas Oncology, El Paso, Texas
  - University of Texas, Houston, Texas
  - Texas Oncology P A Plano East, Plano, Texas
  - Texas Oncology PA Tyler, Tyler, Texas
  - Bon Secours Virginia Health System, Midlothian, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Providence Regional Cancer System, Lacey, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (4):
  - Novartis Investigative Site, Gateshead, New South Wales
  - Novartis Investigative Site, Tiwi, Northern Territory
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
- Canada (7):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (19):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shijiazhuang
  - Novartis Investigative Site, Tianjin
- Germany (27):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Weiden in Der Oberpfalz, Bavaria
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Hildesheim, Lower Saxony
  - Novartis Investigative Site, Bergisch Gladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ravensburg
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Tuenmen
- India (9):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharasthra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bhubaneshwar, Odisha
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Ahmedabad
- Israel (4):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Mexico (3):
  - Novartis Investigative Site, Alc Cuahutemoc, Mexico City
  - Novartis Investigative Site, Tlalpan, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Pan Oncology, Rio Piedras, Puerto Rico
- South Korea (7):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Yangcheon Gu
  - Novartis Investigative Site, Seongnam Gyeonggi
  - Novartis Investigative Site, Seoul
- Taiwan (4):
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (19):
  - Novartis Investigative Site, Sakarya, Adapazari
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Kadikoy
  - Novartis Investigative Site, Izmir, Karsiyaka
  - Novartis Investigative Site, Denizli, Kinikli
  - Novartis Investigative Site, Antalya, Konyaalti
  - Novartis Investigative Site, Istanbul, Sariyer
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Diyarbakır, Sur
  - Novartis Investigative Site, Istanbul, Uskudar
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Adana, Yuregir
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kecioren Ankara
  - Novartis Investigative Site, Konya
  - Novartis Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com